CLINICAL TRIAL: NCT01064323
Title: Global Vascular Effects of Intermittent Pneumatic Compression-Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA00011747
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Coronary Heart Disease
Keywords: intermittent pneumatic leg compression; nitric oxide; vascular endothelial cells; IPC; EECP; atherosclerosis
MeSH Terms: conditions — Coronary Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intermittent leg compression (Other): Intermittent leg compression daily for 3 hrs a day for 4 weeks
  Interventions: Device: Intermittent pneumatic compression of the lower extremities

INTERVENTIONS:
Device: Intermittent pneumatic compression of the lower extremities — IPC will be done for 3 divided hours daily for 4 weeks

SUMMARY:
Intermittent pneumatic compression (IPC) of the lower extremities is a well-established technique for preventing deep vein thrombosis (DVT) and for treating venous stasis. IPC will be done in the home for 3 divided hours every day for 4 weeks. Lab tests, brachial ultrasound and MRI testing will be performed at baseline and after 4 weeks of daily IPC therapy.

See detailed description for increase in healthy control subjects.

DETAILED DESCRIPTION:
Intermittent pneumatic compression (IPC) of the lower extremities is a well-established technique for preventing deep vein thrombosis (DVT) and for treating venous stasis.

Four categories of discoveries suggest that there may be potential of IPC to have global vascular benefits:

1. IPC of the arms prevents DVT in legs;
2. Nitric oxide released by vascular endothelial cells exerts protective effects on blood vessels;
3. IPC increases nitric oxide availability locally in the lower extremity;
4. Nitric oxide may be transported in blood and released at distant sites, particularly in a hypoxic setting. Therefore, we propose to test the effects of lower extremity IPC on global nitric oxide availability.

We will enroll 4 categories of subjects.

The first 3 categories will have only 1 hour of leg compression. Baseline cholesterol will be drawn for screening labs Brachial ultrasound and NO measurements will be done before and after 1 hr of IPC. No MRI will be done on these groups.

Category 4 will have baseline labs and testing to include:

Brachial ultrasound,NO measurements and MRI will be done before and after 4 weeks of daily IPC therapy.

Category 1, 21-40 yrs healthy male or female

Category 2, 50 yrs plus healthy males or females

Category 3, 50 yrs plus aged matched controls with known heart disease

Category 4, 50 yrs plus12 patients with coronary artery disease.

ELIGIBILITY:
Category 1 subjects-healthy volunteers (no MRI required) INCLUSION (N-12) 21 -40 years male or female EXCLUSIONS History of CAD, MI, Cath,CABG,CTA, positive stress test HTN uncontrolled (SBP>140 or DBP>90) DM except diet controlled Cholesterol >200 at screening Smoking last 10 years Acute Medical Illness Inflammatory Phlebitis Infection lower limbs Recent lower limb surgery

Category 2 subjects ( age matched without CAD)(no MRI required) INCLUSION (N-12) 50 plus male or female EXCLUSIONS History of CAD, MI, Cath,CABG,CTA, positive stress test HTN uncontrolled (SBP>140 or DBP>90) DM except diet controlled Cholesterol >200 at screening Smoking last 10 years Acute Medical Illness Inflammatory Phlebitis Infection lower limbs Recent lower limb surgery

Category 3 subjects ( age matched with CAD)(no MRI required) INCLUSION (N-up to 5) 50 plus male or female documented CAD by cath, PTCI, CABG, CTA EXCLUSIONS History of CHF, DVT, PE Angina, active, needing nitrates Acute Medical Illness Inflammatory Phlebitis Infection lower limbs Recent lower limb surgery

Category 4 subjects with MRI (original group) INCLUSIONS(N=12) 50 plus male or female documented CAD by cath, PTCI, CABG, CTA EXCLUSIONS History of CHF, DVT, PE Angina, active, needing nitrates Atrial Fib BMI>35 (MRI) MRI contraindications pregnancy Chronic Inflammatory Disease Acute Medical Illness Inflammatory Phlebitis Infection lower limbs recent lower limb surgery

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Silber, MD, Principal Investigator — JHU
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intermittent Leg Compression: Intermittent leg compression for one hour.
Period: Overall Study
Arm/Group | Intermittent Leg Compression
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
Age, Customized [Count of Participants; unit: Participants]
  24-39 years old | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Brachial Flow Velocity
Description: Brachial flow velocity measured using ultrasound. Units cm/sec.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
cm/sec | 21.0 (6.5)

2. Primary Outcome: Brachial Flow Velocity
Description: Measured using ultrasound, units cm/sec.
Time Frame: 5 minutes into leg intermittent pneumatic compression
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
cm/sec | 18 (6.2)
Statistical Analysis 1: Comparison: Intermittent Leg Compression; Test type: Other — Paired T-test to detect if there was a change from baseline to 5 minutes into intermittent pneumatic compression (IPC); p = 0.02, Paired t-test

3. Primary Outcome: Brachial Flow Velocity
Description: Measured using ultrasound, units cm/sec.
Time Frame: 50 minutes into IPC
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
cm/sec | 17.5 (5.8)

4. Primary Outcome: Brachial Diameter
Description: mm
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
mm | 3.69 (0.70)

5. Primary Outcome: Brachial Diameter
Description: mm
Time Frame: 1 hour after leg IPC
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
mm | 3.67 (0.68)

6. Primary Outcome: Brachial Flow Dilation
Description: Brachial Flow Mediated dilation, mm
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
mm | 0.45 (0.27)

7. Primary Outcome: Brachial Flow Dilation
Description: Brachial Flow Mediated dilation, mm
Time Frame: 1 hour after IPC
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
mm | 3.69 (0.70)

8. Primary Outcome: Brachial Flow Dilation
Description: Brachial Flow Mediated dilation, %
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percentage of dilation
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
percentage of dilation | 13.3 (9.4)

9. Primary Outcome: Brachial Flow Dilation
Description: Brachial Flow Mediated dilation, %
Time Frame: 1 hour after IPC
Measure: Mean (Standard Deviation); unit: percentage of dilation
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
percentage of dilation | 11.5 (7.2)
Statistical Analysis 1: Comparison: Intermittent Leg Compression; Test type: Other; p = 0.2, t-test, 2 sided

10. Primary Outcome: Brachial Occlusion-mediated Constriction
Description: Brachial Occlusion-mediated constriction measured via ultrasound, mm
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
mm | -1.54 (0.51)

11. Primary Outcome: Brachial Occlusion-mediated Constriction
Description: Brachial Occlusion-mediated constriction measured via ultrasound, mm
Time Frame: 1 hour after IPC
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
mm | -1.15 (0.40)

12. Primary Outcome: Brachial Occlusion-mediated Constriction
Description: Brachial Occlusion-mediated constriction measured via ultrasound, %
Time Frame: baseline
Population: Data for this outcome measure was only available for 8 out of 10 participants due to reduced image quality.
Measure: Mean (Standard Deviation); unit: percentage of constriction
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 8
percentage of constriction | -43 (13)

13. Primary Outcome: Brachial Occlusion-mediated Constriction
Description: Brachial Occlusion-mediated constriction measured via ultrasound, %
Time Frame: 1 hour after IPC
Population: Data for this outcome measure was only available for 8 out of 10 participants due to reduced image quality.
Measure: Mean (Standard Deviation); unit: percentage of constriction
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 8
percentage of constriction | -33 (12)

14. Primary Outcome: Plasma Nitrite
Description: nM
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
nM | 112 (26)

15. Primary Outcome: Plasma Nitrite
Description: nM
Time Frame: 1 hour after IPC
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
nM | 90 (15)

16. Primary Outcome: Red Blood Cell Nitric Oxide
Description: nM
Time Frame: baseline
Population: Data was not collected for 1 participant for this outcome measure.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 9
nM | 129 (72)

17. Primary Outcome: Red Blood Cell Nitric Oxide
Description: nM
Time Frame: 1 hour after IPC
Population: Data was not collected for 1 participant for this outcome measure.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 9
nM | 102 (41)

18. Primary Outcome: Plasma S-nitrosothiols
Description: nM
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
nM | 5.79 (4.81)

19. Primary Outcome: Red Blood Cell Nitric Oxide
Description: nM
Time Frame: 1 hour after IPC
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Intermittent Leg Compression
Number analyzed (Participants) | 10
nM | 6.27 (5.79)

ADVERSE EVENTS:
Arm/Group | Intermittent Leg Compression
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes